CLINICAL TRIAL: NCT04564846
Title: A Randomized, Double Blind, Phase 2b Study to Evaluate the Effect of ORMD-0801 Compared to Placebo on Endogenous Glucose Production in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of ORMD-0801 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORA-D-018
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ORMD-0801; Insulin; Fish Oils

STUDY DESIGN:
Intervention Model Description: The subject will receive either placebo or ORMD-0801
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Care Provider, and Investigator will be masked to the intervention (ORMD-0801 or placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be administered a single capsule of placebo( fish oil); placebo will be dispensed and subjects will dose twice a day, once in the morning prior to breakfast and once at night prior to bedtime.
  Interventions: Other: Placebo
- ORMD-0801 (Active Comparator): Subjects will be administered a single 8mg capsule of ORMD-0801; study medication will be dispensed and subjects will dose twice a day, once in the morning prior to breakfast and once at night prior to bedtime.
  Interventions: Drug: ORMD-0801

INTERVENTIONS:
Drug: ORMD-0801 — 8 mg capsules of ORMD-0801 (Oral Insulin)
  Other Names: Oral Insulin
  Arms: ORMD-0801
Other: Placebo — Placebo capsule (Fish Oil)
  Other Names: Fish Oil
  Arms: Placebo

SUMMARY:
This study is designed to explore the efficacy of ORMD-0801 compared to placebo on endogenous glucose production in subjects with type 2 diabetes (T2DM). Subjects will undergo an initial Screening Visit (Visit 0) to establish their eligibility to participate in the study. At Visit 1 (2 weeks after the Screening Visit), qualifying subjects will be randomized to either ORMD-0801 (8 mg) or matching placebo, study medication will be dispensed and subjects will dose, twice a day, once in the morning prior to breakfast and once at night prior to bedtime

DETAILED DESCRIPTION:
This study is designed to explore the efficacy of ORMD-0801 compared to placebo on endogenous glucose production in subjects with type 2 diabetes (T2DM). Subjects will undergo an initial Screening Visit (Visit 0) to establish their eligibility to participate in the study. At Visit 1 (2 weeks after the Screening Visit), qualifying subjects will be randomized to either ORMD-0801 (8 mg) or matching placebo, study medication will be dispensed and subjects will dose, twice a day, once in the morning prior to breakfast and once at night prior to bedtime. Doses will occur at 45 minutes (± 15 minutes) before breakfast and no later than 10 AM each morning, and at 8 PM (± 120 minutes) each night, and no sooner than 1 hour after dinner. Subjects will return to the clinic, 2 weeks later, for Visit 2. At this visit, subject compliance will be assessed, medication will be dispensed, a blood sample will be collected to measure HbA1c and subjects will be questioned for any adverse events. Subjects will be scheduled to return to the clinic in 2 weeks for morning admission (8 AM ± 120 minutes) to the PK unit (Visit 3). Subjects will be provided with standardized meals and the morning dose in-clinic. A light standardized dinner meal will be provided at 6 PM ± 30 minutes. At approximately 8 PM (± 60 minutes, and no sooner than 1 hour after dinner), subjects will be dosed with their study medication and will be started on a 16-hour infusion of [6,6-2H2]-glucose tracer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged, 18 - 70 years.
* Established diagnosis of T2DM for at least 6 months prior to Screening, with HbA1c ≥ 7.5%. and ≤ 11%.
* Stable dose of metformin (at least 1500 mg or maximal tolerated dose) for a period of at least 3 months prior to Screening.
* Taking metformin only or metformin in addition to no more than two of the following: DPP-4, SGLT-2, or TZD.
* Body mass index (BMI) of up to 35 kg/m2 at Screening and stable weight, with no more than 5 kg gain or loss in the 3 months prior to Screening.
* Renal function - eGFR > 30 ml/min/1.73 m2.
* Females of childbearing potential must have a negative serum pregnancy test result at Screening.

Exclusion Criteria:

* Subjects with insulin-dependent diabetes:

  1. Has a history of type 1 diabetes mellitus or a history of ketoacidosis, or subject is assessed by the investigator as possibly having type 1 diabetes mellitus confirmed by a C-peptide < 0.7 ng/mL (0.23 nmol/L).
  2. Has a history of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
* Treatment with glucosidase inhibitor, insulin secretagogues (other than sulfonylureas), glucagon-like peptide 1 (GLP-1) agonists within 3 months prior to Visit 1.
* History of any basal, pre-mix or prandial insulin (greater than 7 days) within 6 months prior to Screening.
* History of > 2 episodes of severe hypoglycemia within 6 months prior to Screening.
* History of hypoglycemic unawareness (episodes of severe hypoglycemia with seizure or requiring third party intervention or documented low blood glucose without associated autonomic symptoms).
* Subjects with the following secondary complications of diabetes:

  1. Active proliferative retinopathy as confirmed by a dilated ophthalmoscopy/retinal photography examination performed (by a qualified person as per the country legislation) within 6 months prior to Screening.
  2. Renal dysfunction: estimated creatinine clearance < 30 ml/min.
  3. History of proliferative retinopathy or severe form of neuropathy or cardiac autonomic neuropathy (CAN).
  4. Uncontrolled or untreated severe hypertension defined as systolic blood pressure above or equal to 180 mmHg and/or diastolic blood pressure above or equal to 120 mmHg.
  5. Presence of unstable angina or myocardial infarction within 6 months prior to Screening, Grade 3 or 4 congestive heart failure (CHF) according to the New York Heart Association (NYHA) criteria, valvular heart disease, cardiac arrhythmia requiring treatment, pulmonary hypertension, cardiac surgery, history/occurrence of coronary angioplasty and/or stroke or transient ischemic attack (TIA) within 6 months prior to Screening.
* Subjects with psychiatric disorders which, per investigator judgment, may have impact on the safety of the subject or interfere with subject's participation or compliance in the study.
* Subjects who needed (in the last 12 months) or may require systemic (oral, intravenous, intramuscular) glucocorticoid therapy for more than 2 weeks during the study period.
* Laboratory abnormalities at Screening including:

  1. C-peptide < 0.7 ng/mL (0.23 nmol/L).
  2. Abnormal serum thyrotropin (TSH) levels below the lower limit of normal or > 1.5X the upper limit of normal.
  3. Elevated liver enzymes (alanine transaminase (ALT), alanine aminotransferase (AST), alkaline phosphatase) > 2X the upper limit of normal.
  4. Very high triglyceride levels (> 600 mg/dL); a single repeat test is allowable.
  5. Any relevant abnormality that would interfere with the efficacy or the safety assessments during study treatment administration.
* Positive history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic hepatitis B or C, primary biliary cirrhosis, or active symptomatic gallbladder disease.
* Positive history of HIV.
* Use of the following medications:

  1. History of any basal, pre-mix or prandial insulin (greater than 7 days) within 6 months prior to Screening.
  2. Administration of thyroid preparations or thyroxine (except in subjects on stable replacement therapy) within 6 weeks prior to Screening.
  3. Administration of systemic long-acting corticosteroids within two months or prolonged use (more than one week) of other systemic corticosteroids or inhaled corticosteroids (if daily dosage is > 1,000 μg equivalent beclomethasone) within 30 days prior to Screening. Intra-articular and/or topical corticosteroids are not considered systemic.
  4. Use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and inhaled steroids (as discussed above), and immunosuppressive or immunomodulating agents.
* Known allergy to soy.
* Subject is on a weight loss program and is not in the maintenance phase, or subject has started weight loss medication (e.g., orlistat or liraglutide), within 8 weeks prior to Screening.
* Subject has had bariatric surgery.
* Subject is pregnant or breast-feeding.
* Subject is a user of recreational or illicit drugs or has had a recent history (within 1 year of Screening) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by > 3 drinks per day or > 14 drinks per week, or binge drinking) at Screening. Occasional intermittent use of cannabinoid products will be allowed provided that no cannabinoid products have been used during the 1 week prior to each visit.
* Subject is smoking more than 10 cigarettes per day.
* One or more contraindications to metformin as per local label.
* History of gastrointestinal disorders (e.g. hypochlorhydria) with the potential to interfere with drug absorption.
* At the Principal Investigator's discretion, any condition or other factor that is deemed unsuitable for subject enrollment into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, M. D., Principal Investigator — Orange County Research Center (OCRC); Ele Ferrannini, M. D., Principal Investigator — CNR Institute of Clinical Physiology
Locations (1):
- Orange County Research Center (OCRC) 14351 Myford Rd., Suite B, Tustin, CA 92780, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gastaldelli A, Baldi S, Pettiti M, Toschi E, Camastra S, Natali A, Landau BR, Ferrannini E. Influence of obesity and type 2 diabetes on gluconeogenesis and glucose output in humans: a quantitative study. Diabetes. 2000 Aug;49(8):1367-73. doi: 10.2337/diabetes.49.8.1367. PMID 10923639
- [Background] Ferrannini E, Gastaldelli A, Iozzo P. Pathophysiology of prediabetes. Med Clin North Am. 2011 Mar;95(2):327-39, vii-viii. doi: 10.1016/j.mcna.2010.11.005. PMID 21281836

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | ORMD-0801
Started | 25 | 24
Completed | 21 | 20
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Principal Investigator requested that the patient withdraw from the study | 1 | 1
Not completed — Subject non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ORMD-0801 | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.19 (6.497) | 58.68 (6.904) | 59.45 (6.742)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 18 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 15 | 23
  Not Hispanic or Latino | 17 | 9 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 13 | 18 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Childbearing Status [Count of Participants; unit: Participants]
  Not Applicable | 18 | 14 | 32
  Of Childbearing Potential | 0 | 0 | 0
  Post Hysterectomy | 3 | 1 | 4
  Surgically Sterilized | 2 | 4 | 6
  At Least one year Post-Menopausal | 2 | 5 | 7
Height [Mean (Standard Deviation); unit: cm] | 170.7 (9.96) | 170.3 (11.50) | 170.5 (10.74)
Weight [Mean (Standard Deviation); unit: Kg] | 88.09 (14.635) | 88.80 (16.546) | 88.438 (15.604)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — BMI = Weight of patient in Kg divided by the square of patient height in meters (meters^2)
  Kg/m^2 | 30.124 (3.5803) | 30.563 (3.7834) | 30.339 (3.6877)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC(0-16)) of Endogenous Glucose Production
Description: The endogenous glucose production in ORMD-0801 and placebo measured by the glucose with tracer attached using AUC(0-16) as the primary parameter. The intravenous infusion of [6,6-2H2]-glucose tracer is administered following administraiton of either placebo or intervention. The pharmacokinetic time points are basline (pre dose), 0.75 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 4 hr, 5 hr, 6 hr, 7 hr, 8 hr, 9 hr, 10 hr, 11 hr, 12 hr, 13 hr, 14 hr, 15 hr, 16 hr post-dose.
Time Frame: Day 28 (1 day)
Population: modified intend-to-treat (mITT) population. mITT consists of all subjects that started on Day 28.
  All 22 mITT placebo subjects came in for Study Day 28. One subject discontinued after the standard blood tests, prior to the pK measurements due to Non-Compliance or Lack of Cooperation. Thus, the sample size on Day 28 for AUC(0-16) is 21, and for the standard blood tests is 22. The 21 subjects that completed Visit 3 (days 28 + 29) were included in this outcome measure.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Placebo | ORMD-0801
Number analyzed (Participants) | 21 | 20
mg*hr/dL | 3436.8 (922.89) | 3139.3 (830.29)
Statistical Analysis 1: Comparison: Placebo vs ORMD-0801; Comparison to Placebo Across All Time Points; Test type: Other; p = 0.1628, Analysis of Covariance; Risk Ratio (RR) = 0.974, 95% CI 2-sided [0.938 to 1.011] — Estimated Difference from Placebo Across All Time Points. Log transformed values analyzed using an Analysis of Covariance model with treatment and time point as effects and baseline HbA1c as a covariate

2. Secondary Outcome: Mean Changes in HbA1c
Description: Mean Changes of HbA1c measured in percentage of glycated hemoglobin
Time Frame: baseline to Day 29 of the treatment period.
Population: modified intent-to-treat population (mITT). The mITT population consists of all subjects that started the Day 28 - 16 hour fast and corresponding measurements.
  All 22 placebo subjects in the mITT population came in for Study Day 28 and started the fast. One subject discontinued prior to the Day 29 measurements due to Non-Compliance or Lack of Cooperation. This is why the Sample Size for Day 28 (and Baseline) is 22 while the Sample Size for Day 29 is 21.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Placebo | ORMD-0801
Number analyzed (Participants) | 22 | 20
percentage of glycated hemoglobin
  Baseline HbA1c | 9.20 (1.214) | 8.51 (1.401)
  Day 29 HbA1c: number analyzed (Participants) | 21 | 20
  Day 29 HbA1c | 9.19 (1.196) | 8.67 (1.319)
  Difference of HbA1c between baseline and Day 29: number analyzed (Participants) | 21 | 20
  Difference of HbA1c between baseline and Day 29 | 0.08 (0.452) | 0.15 (0.637)

3. Secondary Outcome: Area Under the Curve AUC(0-16) of Metabolite Beta-hydroxybutyrate
Description: AUC(0-16) measured in umol*hr/L with blood draws at baseline ( time "0", prior to drug administration), then 45 min, 90 min, 120 min, 150 min, 3-16 hours in one-hour intervals post intervention plus tracer administration via intravenous infusion of [6,6-2H2]-glucose tracer. The AUC measured is AUC(0-16) where "0-16" is 0 pre-dose, 0.75 hr. 1.5 hrs, 2 hrs. 2.5 hrs, 3 hrs, 4 hrs, 5 hrs, 6 hrs, 7 hrs, 8 hrs, 9 hrs, 10 hrs, 11 hrs, 12 hrs, 13 hrs, 14 hrs, 15 hrs, 16 hrs. post dose.
Time Frame: Day 28
Population: modified intend-to-treat (mITT) population. mITT consists of all subjects that started on Day 28.
  All 22 mITT placebo subjects came in for Study Day 28. One subject discontinued after the standard blood tests, prior to the pK measurements due to Non-Compliance or Lack of Cooperation. Thus, the sample size on Day 28 for AUC(0-16) is 21, and for the standard blood tests is 22. The 21 subjects that completed Visit 3 (days 28+ 29) were included in this outcome measure.
Measure: Mean (Standard Deviation); unit: umol*hr/L
Arm/Group | Placebo | ORMD-0801
Number analyzed (Participants) | 21 | 20
umol*hr/L | 3435.8 (3093.36) | 2009.7 (1659.04)
Statistical Analysis 1: Comparison: Placebo vs ORMD-0801; Estimated Difference from Placebo Across All Time Points; Test type: Other; p = 0.0674, Analysis of Covariance; Risk Ratio (RR) = 0.784, 95% CI 2-sided [0.605 to 1.017]; Log transformed values analyzed using an Analysis of Covariance model with treatment and time point as effects and baseline HbA1c as a covariate

4. Secondary Outcome: Area Under the Curve (AUC) of Insulin
Description: The Area Under the Cuve (AUC) measured from baseline (prior to placebo, intervention, and tracer infusion) to sixteen hours post treatment andministration and tracer infusion administration.
  The tracer is [6,6-2H2]-glucose tracer using AUC(0-16). Pharmacokinetic time points are: Baseline (0 hr, pre-dose), then 0.75 hr, 1.5 hrs, 2 hrs, 2.5 hrs., 3 hrs., 4 hrs, 5 hrs, 6 hrs, 7hrs, 8 hrs, 9 hrs, 10 hrs, 11 hrs 12 hrs, 13 hrs, 14 hrs, 15 hrs, 16 hrs (post dose).
Time Frame: Day 28 (one day)
Population: modified intend-to-treat (mITT) population. mITT consists of all subjects that started on Day 28.
  All 22 mITT placebo subjects came in for Study Day 28. One subject discontinued after the standard blood tests, prior to the pK measurements due to Non-Compliance or Lack of Cooperation. Thus, the sample size on Day 28 for AUC(0-16) is 21, and for the standard blood tests is 22. The 21 subjects that completed Visit 3 (days 28+29) were included in this outcome measure.
Measure: Mean (Standard Deviation); unit: uU*hr/mL
Arm/Group | Placebo | ORMD-0801
Number analyzed (Participants) | 21 | 20
uU*hr/mL | 324.8 (147.25) | 425.1 (274.61)
Statistical Analysis 1: Comparison: Placebo vs ORMD-0801; Estimated Difference from Placebo Across All Time Points; Test type: Other — Log transformed values analyzed using an Analysis of Covariance model with treatment and time point as effects and baseline HbA1c as a covariate; p = 0.8182, Analysis of Covariance; Risk Ratio, log = 1.067, 95% CI 2-sided [0.976 to 1.167]

5. Secondary Outcome: Area Under the Curve (AUC) of Free Fatty Acids (FFA)
Description: AUC measured from Baseline (prior to administration of placebo orintervention and to tracer infusion.
  The tracer is [6,6-2H2]-glucose tracer using AUC(0-16). Pharmacokinetic time points are: Baseline (0 hr, pre-dose), then 0.75 hr, 1.5 hrs, 2 hrs, 2.5 hrs., 3 hrs., 4 hrs, 5 hrs, 6 hrs, 7hrs, 8 hrs, 9 hrs, 10 hrs, 11 hrs 12 hrs, 13 hrs, 14 hrs, 15 hrs, 16 hrs (post dose).
Time Frame: Day 28 (one day)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: uEq*hr/L
Arm/Group | Placebo | ORMD-0801
Number analyzed (Participants) | 21 | 20
uEq*hr/L | 7327.2 (1820.31) | 7051.4 (1788.71)
Statistical Analysis 1: Comparison: Placebo vs ORMD-0801; Test type: Other — AUC Parameters analyzed using an Analysis of Covariance model with treatment as the main effect and baseline HbA1c as a covariate; p = 0.8182, Analysis of Covariance; Risk Ratio, log = 1.007, 95% CI 2-sided [0.951 to 1.066]

6. Secondary Outcome: Mean Changes Plasma Glucose Levels
Description: Mean changes in plasma glucose levels measured in mg/dL.
  In this outcome measure, the change from baseline of mean plasma glucose for the placebo arm is calculated as:
  Mean Plasma Glucose (Day 29, 21 subjects) - Mean Plasma Glucose (Baseline, 21 subjects). The Baseline Mean Plasma Glucose based on 21 subjects is 192.7 mg/dL. Therefore, 192.7 mg/dL - 212.3 mg/dL = -19.6 mg./dL
Time Frame: baseline to Day 29 of the treatment period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | ORMD-0801
Number analyzed (Participants) | 22 | 20
mg/dL
  Plasma Glucose at Baseline | 216.4 (55.37) | 187.5 (48.6)
  Plasma Glucose at Day 29: number analyzed (Participants) | 21 | 20
  Plasma Glucose at Day 29 | 192.7 (51.62) | 167.9 (48.58)
  Change in Plasma Glucose from Baseline: number analyzed (Participants) | 21 | 20
  Change in Plasma Glucose from Baseline | -19.6 (46.61) | -19.6 (39.68)
Statistical Analysis 1: Comparison: Placebo vs ORMD-0801; Test type: Other; Parameter analyzed using an Analysis of Variance model with treatment as the main effect; Analysis of Variance = 0.4628

ADVERSE EVENTS:
Time Frame: Baseline (day 0) until discharge/end-of-study day (day 29)
Description: The severity of each AE will be graded according to the NCI CTCAE, version 4.03.
Arm/Group | Placebo | ORMD-0801
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 3/25 | 6/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | ORMD-0801 (N=24)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 3 (3) — Mild
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) — Diarrhoea
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) — Anxiety
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT04564846/Prot_SAP_000.pdf